CLINICAL TRIAL: NCT06868615
Title: AVAVA MIRIA General Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AVAVA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-24-003
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Acne; Acne Scars - Mixed Atrophic and Hypertrophic; Scars; Wrinkle; Pigment; Lesion; Skin Texture Disorder
MeSH Terms: conditions — Acne Vulgaris; Hypertrophy; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): Subjects treated with the AVAVA Device
  Interventions: Device: AVAVA

INTERVENTIONS:
Device: AVAVA — 1550nm Non-Ablative Fractional Laser

SUMMARY:
A general protocol to treat a variety of dermatologic conditions and collect patient feedback.

Primary outcome is the collection and analysis of patient questionnaires related to the overall experience of the device treatment. Secondary outcome measures include physician and subject evaluations in regards to improvement seen in the device as well as assessment of side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 to 70 years of age.
2. Dermatologic condition that can be addressed by the laser, including but not limited to:

   1. Wrinkles
   2. Scars
   3. Acne Scars
   4. Active Acne
   5. Dyschromia
   6. Cutaneous Lesions such as Age or Sun Spots
   7. Melasma
   8. Laxity
3. Willingness to have digital photographs taken of treatment area(s) and agreement with use of photographs for presentation, educational, or marketing purposes.
4. Willingness to comply with the following during the study, including the follow-up period:

   1. maintain consistent skin care regimen on treated areas.
   2. cover treated areas or have very limited sun exposure and, if requested, use an approved sunscreen of SPF 50 or higher.
   3. refrain from using systemic corticosteroids, according to Investigator discretion.
   4. refrain from using topical corticosteroids, retinoids, or prescription skin-lightening medications on the treated areas, according to Investigator discretion.
   5. refrain from any other procedures in the treatment areas.
5. Willingness and ability to comply with study instructions and return for required visits.
6. Subject has read and signed a written informed consent form.
7. Subject lives within 50 miles of study site.
8. Willingness to shave hair in intended treatment area

Exclusion Criteria:

1. Skin pathology or condition that could interfere with evaluation of the study procedure, e.g.,
2. Systemic treatment prescribed within previous 6 months (e.g., oral medication such as isotretinoin)
3. Surgical treatment in the target areas within previous 6 months (e.g., laser surgery)
4. Active vitiligo, psoriasis, or eczema in the treatment area
5. Injection of dermal filler in the target areas within previous 1 month (e.g., collagen, hyaluronic acid filler)
6. Cosmetic procedures in the target areas within prior 3 months (e.g., laser, microdermabrasion, skin peel)
7. Topical treatment applied to target areas within the previous 1 month or according to Investigator discretion.
8. Active suntan and unable or unlikely to refrain from tanning within the follow-up period.
9. Artificial tanning in the target areas within the previous 1 month (e.g., spray, lotion, tanning bed) or intention to use artificial tanning within the follow-up period.
10. Active localized or systemic infection, or an open wound in area being treated.
11. Lesions in the treatment areas suspicious for malignancy (skin cancer, melanoma)
12. History of abnormal wound healing or abnormal scarring (e.g., hypertrophic or keloid)
13. History of connective tissue disease, such as lupus or scleroderma.
14. Any use of medication that is known to increase sensitivity to light according to Investigator's discretion (e.g., topicals that produce sensitivity to light may be used in areas other than the target area).
15. History of gold therapy.
16. History of disease stimulated by heat, such as recurrent herpes simplex or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
17. History of radiation to the treatment area or currently undergoing systemic chemotherapy for the treatment of cancer.
18. For Female: Pregnancy or lactation, or intent to become pregnant within the study period.
19. Significant uncontrolled concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
20. History of immunosuppression/immune deficiency disorder or currently using immunosuppressive medications.
21. Current enrollment in a clinical study of any other unapproved investigational drug or device
22. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect response or participation in this clinical study, or would pose an unacceptable risk to the subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Completion of Post-Treatment Subject Questionnaire | Immediate Post-Treatment
  Post-treatment questionnaire to evaluate the overall patient experience including descriptions of the treatment session and overall patient experience.

SECONDARY OUTCOMES:
Blinded Assessment of Before and After Imaging by Trained Dermatologist | Baseline, 3 Months Post Final Treatment, 6 Months Post Final Treatment, 12 Months Post Final Treatment
  Subject images will be placed in a randomized order and blinded graders will be asked to identify the post-treatment image.
Completion of Follow-Up Subject Questionnaire | 3 Months Post Final Treatment, 6 Months Post Final Treatment, 12 Months Post Final Treatment
  Questionnaire evaluates the subject evaluated results of the study including questions related to the device such as whether or not they would participate in additional treatments or recommend the procedure to friends/family
Physician Rated Satisfaction | Baseline, 3 Months Post Final Treatment, 6 Months Post Final Treatment, 12 Months Post Final Treatment
  Percentage of subject results that treating physician was satisfied with at end of study.
  Physician Rated satisfaction with included options of Very Satisfied, Satisfied, Slightly Satisfied, Neutral, Dissatisfied.
Subject Rated Satisfaction | Baseline, 3 Months Post Final Treatment, 6 Months Post Final Treatment, 12 Months Post Final Treatment
  Percentage of subjects satisfied with their results at end of study. Subject Rated satisfaction with included options of Very Satisfied, Satisfied, Slightly Satisfied, Neutral, Dissatisfied.
Physician Rated Global Clinical Aesthetic Improvement Scale Scoring | Baseline, 3 Months Post Final Treatment, 6 Months Post Final Treatment, 12 Months Post Final Treatment
  Physician will be asked to rate subject improvement on a 5 point scale. 0 - Worsened, 1-No Change, 2-Minor Improvement, 3-Moderate Improvement, 4-Significant Improvement
Subject tolerance of procedure based on pain score during treatment per Visual Analogue Scale | Immediate Post Treatment
  Subjects are asked to rate their pain scores from 0 (No pain) to 10 (worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- AVAVA, Inc., Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual data with other researchers at this time.